CLINICAL TRIAL: NCT05998967
Title: Feasibility and Acceptability of Mobile Mantram Repetition Program for Veterans With PTSD (IVI 22-115)
Brief Title: Pilot Trial of Mobile Mantram Delivery
Acronym: mMRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IVX 23-001; SWIFT-IVI 22-115 (Other Grant/Funding Number: VA SWIFT IVI)
Record Dates: First submitted 2023-08-07; First posted 2023-08-21 (Actual); Results first posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: PTSD
Keywords: Internet-based care; Meditation; Feasibility
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Internet-based instruction in MRP in a self-directed or supported manner
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Self-directed MRP (Experimental): Self-directed instruction in MRP via Internet
  Interventions: Behavioral: Mobile Mantram Repetition Program
- Supported MRP (Active Comparator): Supported instruction in MRP via Internet
  Interventions: Behavioral: Mobile Mantram Repetition Program

INTERVENTIONS:
Behavioral: Mobile Mantram Repetition Program — Internet-based instruction in a meditation practice that involves silent repetition of a spiritual word, one-pointed attention and slowing down
  Other Names: mMRP

SUMMARY:
Mantram Repetition Program (MRP) is a meditation practice that involves silent repetition of a spiritual word, one-pointed attention, and slowing down. It has been shown to help reduce PTSD symptoms among Veterans. This study will look at how Veterans reach to learning MRP via the Internet, either in a self-directed way or with text/phone support.

DETAILED DESCRIPTION:
Easily accessible interventions to address post-traumatic stress disorder (PTSD) can play critical role in reducing PTSD and associated symptoms in Veterans, especially for those who remain symptomatic after treatment with other evidence-based interventions, those who prefer complimentary and integrative therapies, or those who have difficulty accessing traditional face-to-face mental health services. The value of these programs is their ability to provide Veterans with more options in their recovery journey and to reach a broad range of Veterans across multiple settings, including remote rural contexts.

The Mantram Repetition Program (MRP) is a meditation-based practice that consists of the repetition of a spiritual word, one-pointed attention, and slowing down. MRP has been shown to reduce stress in several high-risk populations, and two large randomized, controlled studies show that MRP reduces PTSD symptoms among Veterans. A brief, web-based, self-directed version of MRP has been developed to increase the accessibility of evidence-based PTSD treatment. This version of MRP was tested in a pilot study with undergraduate students, demonstrating its ease of use and success in getting students to engage with the practice. The proposed mixed method study will use the Reach, Effectiveness, Adoption, Implementation, Maintenance (RE-AIM) framework to evaluate the mobile MRP in Veterans with PTSD in two conditions: self-directed and with text/phone support. Data from this pilot study will inform the refinement of the MRP delivery strategy and the development of a full-scale trial to test its effectiveness and implementation outcomes, as well as barriers and facilitators, and other contextual factors.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* Primary clinical complaint of PTSD
* Access to an Internet-enabled device

Exclusion Criteria:

* Cognitive impairment or mental health concerns that necessitated a higher level of care or interfered with ability to engage in study activities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariel J. Lang, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited between December 2021 and August 2022 based on clinical referrals and lists of potential research participants
Pre-assignment Details: Participants had a primary clinical complaint of PTSD and an Internet-enabled device
Period: Overall Study
Arm/Group | Self-directed MRP | Supported MRP
Started | 17 | 19
Completed | 14 | 14
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Self-directed Mantram Repetition Program (MRP): Self-directed instruction in MRP via Internet
  Mobile Mantram Repetition Program: Internet-based instruction in a meditation practice that involves silent repetition of a spiritual word, one-pointed attention and slowing down
- Supported Mantram Repetition Program (MRP): Supported instruction in MRP via Internet
  Mobile Mantram Repetition Program: Internet-based instruction in a meditation practice that involves silent repetition of a spiritual word, one-pointed attention and slowing down
- Total: Total of all reporting groups
Arm/Group | Self-directed Mantram Repetition Program (MRP) | Supported Mantram Repetition Program (MRP) | Total
Number analyzed (Participants) | 17 | 19 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.29 (16.87) | 49.79 (14.52) | 50.50 (15.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 15 | 15 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 13 | 14 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 10 | 11 | 21
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  Vanuatu | 17 | 19 | 36
PTSD Checklist for DSM-5 (PCL-5) [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0-80 with higher scores indicating greater PTSD symptoms.
  units on a scale | 35.94 (18.28) | 30.56 (16.73) | 33.17 (17.46)
Patient Health Questionnaire depression (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0-27 with higher scores indicating greater depression.
  units on a scale | 11.47 (6.32) | 10.58 (5.58) | 11.00 (5.87)
Insomnia Severity Index (ISI) [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0-28 with higher scores indicating greater insomnia.
  units on a scale | 15.94 (6.55) | 13.00 (8.13) | 14.39 (7.47)

OUTCOME MEASURES:

1. Primary Outcome: Eligibility Rate
Description: Rate of eligibility among those screened for participation
Time Frame: Day 0
Population: Screened individuals
Measure: Count of Participants; unit: Participants
Groups:
- Total Enrolled Sample: All Veterans screened for participation in the study
Arm/Group | Total Enrolled Sample
Number analyzed (Participants) | 59
Participants | 38

2. Primary Outcome: Initiation Rate
Description: Rate of intervention initiation among eligible Veterans
Time Frame: Day 1
Population: Eligible individuals
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Veterans: Number of individuals meeting all eligibility requirements
Arm/Group | Eligible Veterans
Number analyzed (Participants) | 38
Participants | 36

3. Primary Outcome: Completion Rate
Description: Rate of intervention completion among eligible Veterans
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Eligible Veterans
Number analyzed (Participants) | 38
Participants | 28

4. Primary Outcome: Credibility
Description: Average Veteran perception of the logic, utility and expected benefit of treatment rated on a scale of 0 (not at all) to 8 (very)
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-directed MRP | Supported MRP
Number analyzed (Participants) | 17 | 19
units on a scale | 4.78 (1.35) | 5.23 (1.65)

5. Primary Outcome: Abbreviated Client Satisfaction Questionnaire (CSQ-8)
Description: Degree of satisfaction with care received as measured by 4 items from the CSQ-8, creating a 4-item total score. Scores range from 4-16 with higher scores indicating greater satisfaction.
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Self-directed MRP | Supported MRP
Number analyzed (Participants) | 14 | 14
score on a scale | 11.75 (3.41) | 12.92 (2.29)

6. Primary Outcome: Acceptability of Intervention Measure (AIM)
Description: Perceived acceptability of the intervention as measured by an AIM average score. Scores range from 1-5 with higher scores indicating greater acceptability.
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-directed MRP | Supported MRP
Number analyzed (Participants) | 14 | 14
units on a scale | 4.46 (0.59) | 4.23 (0.81)

7. Primary Outcome: Intervention Appropriateness Measure (IAM)
Description: Perceived appropriateness of the intervention as measured by an IAM average score. Scores range from 1-5 with higher scores indicating greater appropriateness.
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-directed MRP | Supported MRP
Number analyzed (Participants) | 14 | 14
units on a scale | 3.54 (1.05) | 3.81 (0.80)

8. Primary Outcome: Feasibility of Intervention Measure (FIM)
Description: Perceived feasibility of the intervention as measured by an FIM average score. Scores range from 1-5 with higher scores indicating greater feasibility.
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-directed MRP | Supported MRP
Number analyzed (Participants) | 14 | 14
units on a scale | 4.12 (0.48) | 3.77 (0.90)

9. Secondary Outcome: Mantram Practice
Description: Frequency of mantram practice in the past week as 0-7 days
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: days/week
Arm/Group | Self-directed MRP | Supported MRP
Number analyzed (Participants) | 14 | 14
days/week | 4.93 (2.34) | 5.00 (1.75)

10. Secondary Outcome: PTSD Checklist for DSM-5 (PCL-5)
Description: PTSD symptoms at post-treatment as measured by the PCL-5 total score. Scores range from 0-80 with higher scores indicating greater PTSD symptoms.
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Self-directed MRP | Supported MRP
Number analyzed (Participants) | 14 | 14
score on a scale | 31.00 (21.45) | 27.71 (19.23)

11. Secondary Outcome: Patient Health Questionnaire Depression Items (PHQ-9)
Description: Depression at post-treatment as measured by the PHQ-9 total score. Scores range from 0-27 with higher scores indicating greater depression.
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Self-directed MRP | Supported MRP
Number analyzed (Participants) | 14 | 14
score on a scale | 11.50 (8.13) | 9.86 (6.56)

12. Secondary Outcome: Insomnia Severity Index
Description: Insomnia at post-treatment as measured by the ISI total score. Scores range from 0-28 with higher scores indicating greater insomnia.
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Self-directed MRP | Supported MRP
Number analyzed (Participants) | 14 | 14
score on a scale | 15.79 (7.64) | 12.14 (8.17)

ADVERSE EVENTS:
Time Frame: 4 week study period
Arm/Group | Self-directed MRP | Supported MRP
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/19
Other Adverse Events (participants affected / at risk) | 0/17 | 1/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Self-directed MRP (N=17) | Supported MRP (N=19)
Emotional distress (Psychiatric disorders) | 0 (0) | 1 (1) — Distress related to assessment of mental health symptoms

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/67/NCT05998967/Prot_SAP_001.pdf
  • Informed Consent Form (2023-05-18): https://cdn.clinicaltrials.gov/large-docs/67/NCT05998967/ICF_000.pdf